CLINICAL TRIAL: NCT01126398
Title: The Role of Patient Expectations in Traumatic Orthopedic Outcomes: the Development of the Trauma Expectation Factor Trauma Outcome Measure (TEFTOM)
Brief Title: Trauma Expectation Factor Trauma Outcome Measure
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: TEFTOM
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2010-05

CONDITIONS: Ankle Fracture; Pilon Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ankle / dist. tibia fracture fixation
  Interventions: Procedure: ankle or distal tibia surgery

INTERVENTIONS:
Procedure: ankle or distal tibia surgery — internal fixation for ankle or distal tibia fracture

SUMMARY:
This study is designed as a prediction trial. That is, our primary purpose is to develop a model that can be applied clinically as a user-friendly "baseline" questionnaire that is capable of predicting "success" or "failure" based on a patient's pre-surgical expectations of their final outcome. In the process, a secondary goal is to develop an outcomes measure.

DETAILED DESCRIPTION:
Aims:

1. To develop a novel, psychometrically sound, trauma patient expectation instrument that: a) demonstrates content validity; b) considers patient and surgeon expectations; c) predicts orthopedic outcomes; d) is reliable; e) is patient friendly; and f) is easy to score and interpret. This will be known as the Trauma Expectation Factor (TEF).
2. To develop a novel, psychometrically sound, trauma patient outcomes instrument that: a) demonstrates content validity; b) measures current condition in the same domains as the expectation instrument; c) demonstrates construct validity; d) demonstrates criterion validity; e) is reliable; f) is patient friendly; and g) is easy to score and interpret. This will be known as the Trauma Outcomes Measure (TOM).

Hypotheses:

H#1. A simple pre-surgical questionnaire that measures patient expectations (i.e., Trauma Expectation Factor) after an ankle fracture requiring surgery will predict an "expected" score on a standardized disease-specific ankle instrument (i.e., AAOS Foot and Ankle Core Score).

H#2. A similar instrument that is reworded to assess current condition (i.e., Trauma Outcomes Measure) instead of expectations, is a valid, reliable, and responsive measure of a traumatic patient's condition.

H#3. Patient and surgeon expectations of final outcome status are different; however, the differences get smaller over time.

ELIGIBILITY:
Inclusion Criteria:

* Isolated ankle or distal tibia fracture
* Scheduled for and undergoing surgery for their fracture
* 18 years of age or older

Exclusion Criteria:

* Subject has previously undergone internal fixation surgery for this ankle fracture
* Subject has disease entity, or condition that precludes likelihood of bony union (eg, metastatic cancer, metabolic bone disease)
* Subject has severe dementia or other severe mental health problem that may preclude him/her from completing study questionnaires
* Subject is participating in other competing clinical research that may interfere with participation in this research
* Subject is unlikely to attend study related follow-up visits
* Subject has polytrauma (more than one organ system compromised)
* Subject has fracture(s) other than ankle fracture
* Subject is a prisoner
* Fracture occurred more than 4 weeks ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who expericenced an ankle or pilon fracture presenting to the emergency room or orthopedic department were asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
patient reported outcomes | 12 months post-op
  The patient reported outcome includes the Trauma Outcome Measure (TOM), the AAOS Foot and Ankle Core Score, the Foot and Ankle Outcome Scores (FAOS), a 10mm visual analogue scale (VAS), and the SF-36.

SECONDARY OUTCOMES:
Clinician based outcomes | 12 months post-op
  Bony union was assessed using X-Rays.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Suk, Professor, Principal Investigator — Orthopaedic Trauma Service, Universitiy of Florida - Shands Jacksonville
Locations (5):
- United States (3):
  - Orthopedic Trauma Service, University of Florida - Shands Jacksonville, Jacksonville, Florida
  - Department of Orthopaedic Surgery, Hospital for Special Surgery, New York, New York, New York
  - Department of Orthopaedic Surgery, New York Presbyterian Hospital, New York, New York, New York
- Department of Orthopedic Surgery, Ribeirao Preto Medical School - University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil
- Department of Orthopaedic Trauma, Foothills Medical Center, Calgary, Calgary, Alberta, Canada